CLINICAL TRIAL: NCT04591925
Title: Open, Controlled, and Randomized Cross-Over Pilot Study of an Investigational Extended Wear Insulin Infusion Set During Home Use in People With Type 1 Diabetes Mellitus
Brief Title: SteadiSet™ Pilot Study (SteP Study)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim analysis
Sponsor: Capillary Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 150-1139-00
Record Dates: First submitted 2020-10-02; First posted 2020-10-19 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Diabetes Mellitus, Type I; IDDM; Diabetes Mellitus, Insulin-Dependent, 1; Type 1 Diabetes; Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Investigative Device - SteadiSet™" device with coil-reinforced soft polymer indwelling cannula (Experimental): Participants are randomized into the investigational device (SteadiSet™) insulin infusion set group and then switched to a Commercially available infusion set (using a soft Teflon indwelling cannula) group. At the Day of Insertion (Day 0) clinic visit, study participants will insert (under supervision) the investigational infusion set. Upon completion of a wear period (after 14 days or sooner, in the event that infusion set change out has occurred), participants will be asked to insert a new set at home and thus start the next 14-day wear period. After two periods participants will return to the study site to cross over into the last two periods with the Control device infusion set. A total of four infusion sets will be studied in each participant, two Investigational Device infusion sets and two commercially available Teflon infusion sets.
  Interventions: Device: Investigative insulin infusion devcie
- Commercially available Insulin Infusion device using a soft Teflon indwelling cannula (Active Comparator): Participants are randomized into the Commercially available insulin infusion set (using a soft Teflon indwelling cannula) group and then switched to Investigative Device infusion set (SteadiSet™) group. At the Day of Insertion (Day 0) clinic visit, study participants will insert (under supervision) the Control infusion set. Upon completion of a wear period (after 14 days or sooner, in the event that infusion set change out has occurred), participants will be asked to insert a new set at home and thus start the next 14-day wear period. After two periods participants will return to the study site to cross over into the last two periods with the Investigational Device infusion set. A total of four infusion sets will be studied in each participant, two Investigational Device infusion sets and two commercially available Teflon infusion sets.
  Interventions: Device: Control Device insulin infusion devcie

INTERVENTIONS:
Device: Control Device insulin infusion devcie — Control Device - Commercially available insulin infusion device using a soft Teflon indwelling cannula
  Arms: Commercially available Insulin Infusion device using a soft Teflon indwelling cannula
Device: Investigative insulin infusion devcie — Investigative insulin infusion device with coil-reinforced soft polymer indwelling cannula
  Arms: Investigative Device - SteadiSet™" device with coil-reinforced soft polymer indwelling cannula

SUMMARY:
This study will evaluate the safety and effectiveness of how well blood glucose is managed when a participate wears the investigational SteadiSet™ Infusion Set (SteadiSet device) for up to 14 days post-insertion when compared to a Teflon Control infusion set.

DETAILED DESCRIPTION:
Up to 48 adult participants, ages 18-70, diagnosed with type 1 diabetes mellitus (T1DM) may be enrolled, aiming for approximately 40 completers. Participants must have ≥6 months experience using a rapid-acting insulin analog delivered via tubing-based insulin pumps and infusion sets and must demonstrate willingness and ability to use a continuous glucose monitor (CGM). Study participants will be drawn from existing T1DM patient populations meeting the study eligibility at the study center.

Existing patient populations at the study center will be screened for study eligibility within 21 days of planned study randomization. Eligible participants will complete written informed consent and will be assigned a unique study ID. Enrolled participants will complete a one-week run-in period to assess participant compliance to collect adequate CGM data (>80% of possible readings) with the study CGM. Participants who do not achieve this goal will be given a second week of CGM data collection; failing the second week of adequate data collection they will be discontinued from study.

At the Day of Insertion (Day 0) clinic visit, study participants will be randomized to insert (under supervision) either an investigational SteadiSet or a commercially-available Teflon infusion set (different to their routine set); an automatic insertion device will be used for all infusion set insertion procedures during study. Participants will undergo training and be provided written instructions if infusion set failure occurs and set change is required during the up to 14-day wear period. Visual inspection and photographic documentation of the infusion set insertion site will be recorded at Day 0. Participants will be asked to conduct daily insertion site visual inspection and report/record site reactions, unexplained hypo- and hyperglycemic events and symptoms and/or the need for infusion set change (Days +1 to +14).

Upon completion of a wear period (after 14 days or sooner, in the event that infusion set change out has occurred), participants will be asked to insert a new set at home and thus start the next 14-day wear period. After two periods participants will return to the study site to cross over into the last two periods with the respective other infusion set (SteadiSet or Control device, self-insertion under supervision). A total of four infusion sets will be studied in each participant, two SteadiSet and two commercially available Teflon infusion sets.

Insulin therapy will be performed by the participants using their own insulin pump as under routine conditions. Participants will continue to use the rapid acting insulin analog they also use under routine conditions (insulins aspart or lispro). Insulin reservoir and tubing change will be performed as under routine conditions every 6 (insulin aspart) or 7 (insulin lispro) days (or sooner for participants who use more than 300 units every 6-7 days). The infusion set will NOT be changed at the time of reservoir change.

Continuous glucose monitoring will be performed throughout the study. At least four-point capillary blood glucose measurements will be performed each day (pre-meal, bed-time). Participants will be asked to perform capillary ketone measurements in case of unexplained hyperglycemia (glucose >250 mg/dL or 14 mmol/L). Unexplained hypo- or hyperglycemia measured by CGM needs to be verified by capillary glucose measurements. Data from the participant's blood glucose and ketone monitor will be downloaded upon completion of each infusion set wear period. The diary will be collected at each study center visit.

End-of-study will occur at the clinic visit following the fourth study period or upon 30-day follow-up of ongoing adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Participants are 18 - 70 years of age, both inclusive
* Participant is in generally good health, as determined by the investigator
* Participant is willing and able to individually complete written informed consent and agrees to comply with all study related testing and examinations
* Participant must be geographically stable (e.g., expects to be available and capable of returning for all study specified test and examinations) during the study period
* Participant has been diagnosed with T1DM for at least 12 months
* C-peptide <0.6 nmol/L at screening
* Participant can provide a minimum of 14 days of insulin pump data to demonstrate pump use compliance
* Participant is willing to perform serum ketone measurements whenever the blood glucose is determined to be greater than 250 mg/dL (14 mmol/L) using a ketone meter and strips provided by the sponsor
* Participant has BMI in the range 18 - 35 kg/m2, both inclusive
* Participant has experience infusing insulin lispro or aspart for at least 6 months
* Participant has been using an insulin pump with commercially available infusion sets for at least 6 months
* Participant shows willingness to use CGM and successfully completes at least 1 week of successful trial with the Dexcom G6 (readings for at least 80% of the time can be retrieved)
* Participant has ability to understand and comply with protocol procedures and to provide informed consent

Exclusion Criteria:

* Participants routinely using steel insulin infusion sets who due to medical/skin conditions cannot switch to a Teflon set in the control ar
* Participants whose average total daily insulin dose exceeds 85 units/day (i.e. typically change insulin reservoirs more often than every 3.5 days on average
* Participants using any other medication than insulin to control their diabetes
* Participants who routinely change their commercial insulin infusion sets twice weekly or less often (wear time > 3.5 days)
* Female participant is pregnant, planning to become pregnant, not using adequate method of contraception or nursing
* Participant has abnormal skin at intended device infusion sites (existing infection, inflammation, burns, or other extensive scarring)
* Participant has HbA1C > 9.0% at screening
* Participant has documented history in last 6 months of severe hypoglycemia associated with cognitive dysfunction sufficiently severe to require third party intervention or a history of impaired awareness of hypoglycemia.
* Participant has a history of diabetic ketoacidosis in the last 6 months
* Participant has known cardiovascular disease considered to be clinically relevant by the investigator
* Participant has known arrhythmias considered to be clinically relevant by the investigator
* Participant has known history of: Cushing's Disease, pancreatic islet cell tumor, or insulinoma
* Participant has: Lipodystrophy, extensive lipohypertrophy, as assessed by the investigator
* Participant is undergoing current treatment with: Systemic oral or intravenous corticosteroids, monoamine oxidase (MAO) inhibitors, non-selective beta-blockers, growth hormone, thyroid hormones, unless use has been stable during the past 3 months
* Participant has significant history of any of the following, that in the opinion of the investigator would compromise the participant's safety or successful study participation: Alcoholism, drug abuse
* Significant acute or chronic illness, that in the investigator's opinion, might interfere with participant safety or integrity of study results
* Planned operation, MRI or CT which require removal of infusion set or CGM sensor during wear periods
* Current participation in another clinical drug or device study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2021-11-02 (Actual)

PRIMARY OUTCOMES:
Days of successful insulin delivery through the SteadiSet™ insulin infusion device versus a commercially available insulin infusion set | up to 14 days
  Successful insulin delivery period is defined as the days from infusion set insertion to either a removal of the infusion set due to normal use or removal of the infusion set due to set failure. a removal due to normal use or an infusion set failure, defined as:
  * The occurrence of hyperglycemia (glucose >250 mg/dL or 14 mmol/L), not responsive to a pump bolus dose where response to the bolus is defined as a fall of at least 50 mg/dL or 2.8 mmol/L in blood glucose within one hour
  * The occurrence of any hyperglycemic episode (glucose > 250 mg/dL or 14 mmol/L) not associated with acute intercurrent illness, but with a concurrent ketone level ≥0.6 mmol/L, or
  * Signs of infection at the infusion site (e.g. erythema or induration >1 cm in diameter) at the investigator's discretion, or
  * Occurrence of a non-resolvable insulin pump occlusion alarm signal

CONTACTS AND LOCATIONS:
Overall Officials: Julia Mader, Professor, Principal Investigator — Medical University of Graz
Locations (1):
- Medizinische Universität Graz, Graz, Austria